CLINICAL TRIAL: NCT04147195
Title: NASH EXploratory Single and COmbination Treatment (NEXSCOT): An Open Label, Multicenter, Platform Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Various Single and Combination Treatments in Patients With Non-alcoholic Fatty Liver Disease (NAFLD) Who Manifest a Non-alcoholic Steatohepatitis (NASH)-Like Biomarker Phenotype
Brief Title: Study of Various Treatments in Non-alcoholic Fatty Liver Disease (NAFLD) Patients Who Have Aspects of Non-alcoholic Steatohepatitis (NASH)
Acronym: NEXSCOT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CADPT02A12001; 2018-002692-17 (EudraCT Number)
Record Dates: First submitted 2019-10-22; First posted 2019-11-01 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Non-alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: Non-alcoholic fatty liver disease; NAFLD; Non-alcoholic steatohepatitis; NASH; Platform design; LYS006; LJN452; Tropifexor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — tropifexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYS006 (Experimental): LYS006 20 mg was administered orally twice per day (b.i.d) for 12 weeks
  Interventions: Drug: LYS006
- LYS006 + LJN452 (Experimental): LYS006 20 mg was administered orally twice per day (b.i.d) in addition to LJN452 200ug administered orally once daily for 12 weeks
  Interventions: Drug: Tropifexor

INTERVENTIONS:
Drug: LYS006 — 5 mg LYS006 capsules orally administered 20 mg b.i.d for 12 weeks
  Arms: LYS006
Drug: Tropifexor — 100 ug LJN452 capsules orally administered 200ug once daily for 12 weeks
  Other Names: LJN452
  Arms: LYS006 + LJN452

SUMMARY:
This clinical study was designed to evaluate the safety, tolerability, pharmacokinetics and efficacy of various single and combination treatments in adult patients with non-alcoholic fatty liver disease (NAFLD) who manifest a non-alcoholic steatohepatitis (NASH)-like biomarker phenotype.

DETAILED DESCRIPTION:
This was a Phase II, non-confirmatory, multicenter, open label, platform study in NAFLD participants with a NASH-like biomarker phenotype to examine the effects of single and combination therapies over 12 weeks of treatment. The study consisted of four distinct study periods:

* Screening Period (Day -60 to -28): Lasted up to a maximum of 33 days where participants were assessed for inclusion and exclusion criteria prior the baseline assessments.
* Baseline Period (Day -27 to -1): Lasted up to a maximum of 27 days and comprised baseline assessments and randomization.
* Treatment Period (Day 1 to 85): Participants were randomized in a 1:1 ratio to LYS006 20 mg (twice a day) arm or to LYS006 20 mg (twice a day) and tropifexor 200ug (once a day). Participants were treated daily during 12 weeks.
* Follow-up Period (Day 85 to 113): After completion of the treatment period, participants were observed until the End Of Study (EOS) visit at Day 113.

ELIGIBILITY:
Inclusion Criteria:

Phenotypic diagnosis of NASH based on the presence of all of the following:

* ALT ≥ 43 IU/L (males) or ≥ 28 IU/L (females)
* BMI ≥ 27 kg/m2 (race other than Asian) or ≥ 23 kg/m2 (Asian race)
* History of type 2 diabetes mellitus with HbA1c ≤ 9%
* ELF test score ≥ 8.5 and ≤ 10.5
* Liver fat ≥ 8%
* Patients must weigh between 40 kg (88 lbs.) and 150 kg (330 lbs.)

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of randomization or within 3 months, whichever is longer
* Use of obeticholic acid (OCA) or pharmacologically-active weight loss drugs within 1 month of randomization
* Use of strong CYP3A4/5 inhibitors or strong CYP3A4 inducers within 5 half-lives or 7 days of randomization, whichever is longer
* History or presence of other concomitant liver diseases
* History or current diagnosis of ECG abnormalities
* Patients with contraindications to MRI imaging
* Current or history of significant alcohol consumption
* Clinical evidence of hepatic decompensation or severe liver impairment
* Women of child bearing potential (unless on highly effective methods of contraception)
* Presence of liver cirrhosis
* Use of OAT3 inhibitors within 5 half-lives or 7 days of randomization, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (8):
  - Novartis Investigative Site, Coronado, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, South Bend, Indiana
  - Novartis Investigative Site, Morehead City, North Carolina
  - Novartis Investigative Site, San Antonio, Texas
- Novartis Investigative Site, Buenos Aires, Argentina
- Novartis Investigative Site, Essen, Nordrhine Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Frias J, Schmouder R, Lawitz E, Zhang Y, Zhou H, Badman MK, Ukomadu C, Weiss HM, Zack J, Yadav B, Martic M, Drakeford C, Koo P, Naoumov NV, Greenbaum LE. Clinical trial: A Phase 2 Randomised Platform Study to Assess Monotherapy and Combination Treatment Regimens in Metabolic Dysfunction-Associated Steatohepatitis. Aliment Pharmacol Ther. 2025 Nov 26. doi: 10.1111/apt.70475. Online ahead of print. PMID 41305844
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 sites in 3 countries.
Pre-assignment Details: Participants underwent a Screening period of up to 33 days followed by a Baseline assessment period of up to 27 days.
Period: Overall Study
Arm/Group | LYS006 | LYS006 + LJN452
Started | 20 | 21
PD Analysis Set (Participants with available PD data and no major protocol deviations with impact on PD data.) | 20 | 17
Completed | 16 | 15
Not Completed | 4 | 6
Not completed — Adverse Event | 0 | 3
Not completed — Study Terminated by Sponsor | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYS006 | LYS006 + LJN452 | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: Year] | 52.0 (9.23) | 54.9 (8.36) | 53.5 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 19 | 17 | 36
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs including significant changes from baseline in vital signs, electrocardiograms and laboratory parameters qualifying and reported as AEs. The number of participants in each category is reported in the table.
Time Frame: From the start of treatment to 28 days after end of treatment, assessed up to maximum duration of 113 Days
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 21
Participants
  AEs | 14 | 17
  Treatment-related AEs | 2 | 15
  SAEs | 0 | 0
  AEs leading to discontinuation of study treatment | 0 | 3

2. Secondary Outcome: Change From Baseline in Non-invasive Markers of Hepatic Fibrosis: Enhanced Liver Fibrosis Test (ELF) Score
Description: The markers of fibrosis assessed in this test comprised hyaluronic acid (HA), tissue inhibitor of metalloproteinase (TIMP1) and procollagen III N-terminal peptide (PIIINP); these are components of the extracellular matrix and basement sinusoidal membrane of the liver and are elevated during fibrogenesis as a result of activation of the hepatic stellate cell. The ELF test is a composite score: < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates decreased fibrosis.
Time Frame: Baseline and Days 57, 85 and EOS (Day 113)
Population: The overall number of participants analyzed includes all participants in the PD analysis set. The number analyzed per row represents participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
Scores on a scale
  Day 57: number analyzed (Participants) | 17 | 12
  Day 57 | -0.25 (0.564) | 0.29 (0.286)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | -0.12 (0.780) | 0.18 (0.687)
  EOS: number analyzed (Participants) | 13 | 11
  EOS | 0.01 (0.713) | 0.09 (0.461)

3. Secondary Outcome: Change From Baseline in Cholesterol: Fasting Lipid Profile Endpoint
Description: Fasting lipid profile (total cholesterol) was examined as a cardiometabolic risk parameter. Total cholesterol was measured on blood samples under fasted conditions and analyzed at a central laboratory.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates cardiovascular risk.
Time Frame: Baseline and Days 15, 29, 43, 57, 85 and EOS (Day 113)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
mmol / L
  Day 15: number analyzed (Participants) | 19 | 17
  Day 15 | -0.025 (0.5814) | 0.086 (0.8825)
  Day 29: number analyzed (Participants) | 18 | 15
  Day 29 | -0.058 (0.6058) | 0.431 (1.0688)
  Day 43: number analyzed (Participants) | 16 | 14
  Day 43 | -0.109 (0.6758) | 0.474 (1.0364)
  Day 57: number analyzed (Participants) | 17 | 12
  Day 57 | -0.246 (0.6341) | 0.463 (1.3026)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | 0.001 (0.8558) | 0.754 (0.9915)
  EOS: number analyzed (Participants) | 14 | 11
  EOS | -0.283 (1.1182) | 0.249 (0.5175)

4. Secondary Outcome: Change From Baseline in Percent Liver Fat at Day 85
Description: Percent (%) Liver fat was measured by Magnetic Resonance Imaging Proton Density Liver Fat Fraction (MRIPDFF). Participants underwent magnetic resonance imaging twice during the course of the study (baseline and end of treatment) to quantitate liver fat.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates a reduction in a component of NAFLD.
Time Frame: Baseline and Day 85
Population: The overall number of participants analyzed includes all participants in the PD analysis set with evaluable data for the endpoint.
Measure: Mean (Standard Deviation); unit: Percentage of Liver Fat
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 14 | 11
Percentage of Liver Fat | -3.74 (3.470) | -7.52 (5.846)

5. Secondary Outcome: Change From Baseline in Total Body Weight
Description: Body weight (to the nearest 0.1 kilogram [kg] was measured on a calibrated scale. The measurement was performed with the study participant in underwear and without shoes; or while wearing minimal indoor clothing.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates improvement in obesity.
Time Frame: Baseline and Days 15, 29, 43, 57, 85 and EOS (Day 113)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
kg
  Day 15: number analyzed (Participants) | 19 | 17
  Day 15 | -0.21 (1.412) | -1.09 (2.030)
  Day 29: number analyzed (Participants) | 18 | 15
  Day 29 | -0.27 (1.513) | -1.17 (2.455)
  Day 43: number analyzed (Participants) | 16 | 14
  Day 43 | -0.24 (1.664) | -1.94 (2.780)
  Day 57: number analyzed (Participants) | 17 | 12
  Day 57 | -0.48 (1.548) | -2.97 (3.144)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | -0.54 (2.334) | -3.33 (2.892)
  EOS: number analyzed (Participants) | 14 | 11
  EOS | 0.17 (2.753) | -2.56 (2.789)

6. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) at Day 85
Description: HOMA-IR is a test that uses a simultaneous fasting blood glucose test and fasting insulin test to accurately estimate the degree of insulin resistance (IR) and β-cell function (the cells of the pancreas that produce insulin). HOMA-IR scores are classified as follows: Insulin sensitive is considered less than 1.0, Healthy is considered 0.5-1.4, Above 1.8 is early insulin resistance and Above 2.7 is considered significant insulin resistance
  HOMA-IR= [Fasting glucose (mmol/L) x (fasting insulin (pmol/L)/6)] / 22.5
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates improvement in insulin sensitivity.
Time Frame: Baseline and Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 14 | 9
HOMA-IR score | -3.74 (9.865) | 1.67 (7.741)

7. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Fasting Glucose was examined as a cardiometabolic risk parameter. Total fasting glucose was measured on blood samples under fasted conditions and analyzed at a central laboratory.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates improvement in glycemic control.
Time Frame: Baseline and Days 15, 29, 43, 57, 85 and EOS (Day 113)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
mmol / L
  Day 15: number analyzed (Participants) | 19 | 17
  Day 15 | 0.26 (2.609) | 0.26 (2.402)
  Day 29: number analyzed (Participants) | 18 | 15
  Day 29 | -0.04 (3.541) | 0.61 (2.362)
  Day 43: number analyzed (Participants) | 15 | 14
  Day 43 | -0.53 (3.655) | 1.05 (2.449)
  Day 57: number analyzed (Participants) | 17 | 12
  Day 57 | -0.82 (3.176) | 0.84 (1.960)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | -1.74 (3.810) | 0.41 (2.023)
  EOS: number analyzed (Participants) | 14 | 11
  EOS | -1.01 (3.627) | -0.40 (1.563)

8. Secondary Outcome: Change From Baseline in Fasting Insulin at Day 85
Description: Fasting insulin was examined as a cardiometabolic risk parameter. Total fasting insulin was measured on blood samples under fasted conditions and analyzed at a central laboratory.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates improvement in insulin sensitivity.
Time Frame: Baseline and Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol / L
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 14 | 9
pmol / L | -28.36 (139.23) | 14.23 (63.875)

9. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c was examined as a cardiometabolic risk parameter. HbA1c was measured on blood samples under fasted conditions and analyzed at a central laboratory.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates improvement in glycemic control.
Time Frame: Baseline and Days 15, 29, 43, 57, 85 and EOS (Day 113)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
Percentage
  Day 15: number analyzed (Participants) | 18 | 17
  Day 15 | 0.10 (0.194) | 0.08 (0.338)
  Day 29: number analyzed (Participants) | 18 | 15
  Day 29 | 0.03 (0.431) | 0.21 (0.487)
  Day 43: number analyzed (Participants) | 16 | 14
  Day 43 | -0.02 (0.544) | 0.31 (0.884)
  Day 57: number analyzed (Participants) | 17 | 11
  Day 57 | -0.11 (0.730) | 0.36 (0.680)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | -0.48 (0.834) | -0.03 (0.863)
  EOS: number analyzed (Participants) | 14 | 11
  EOS | -0.59 (0.961) | 0.34 (0.359)

10. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: Alanine aminotransferase (ALT) is an enzyme found primarily in the liver. ALT is increased with liver damage. In this study, the blood levels of ALT was used to detect liver inflammation.
  Baseline is defined as the mean of the last 2 non-missing measurements taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates a reduction in liver inflammation.
Time Frame: Baseline and days 15, 29, 43, 57, 85 and EOS (Day 113)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U / L
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
U / L
  Day 15: number analyzed (Participants) | 19 | 16
  Day 15 | 0.97 (18.255) | -19.75 (25.617)
  Day 29: number analyzed (Participants) | 18 | 15
  Day 29 | -6.92 (22.166) | -9.63 (13.774)
  Day 43: number analyzed (Participants) | 16 | 14
  Day 43 | -11.13 (21.624) | -8.68 (14.573)
  Day 57: number analyzed (Participants) | 17 | 12
  Day 57 | -12.09 (25.401) | -17.04 (12.841)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | -7.21 (34.702) | -11.14 (26.318)
  EOS: number analyzed (Participants) | 14 | 11
  EOS | -14.50 (29.619) | -8.05 (14.570)

11. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP)
Description: High-sensitivity C-reactive protein is a blood test marker for inflammation in the body. HsCRP was measured from a blood sample and analyzed at a central laboratory.
  Baseline is defined as the last non-missing measurement taken at the Screening and Baseline visits (prior to the first dose of study drug administered at the Day 1). A negative change from Baseline indicates a reduction in liver inflammation.
Time Frame: Baseline and Days 57, 85 and EOS (Day 113)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg / L
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 17
mg / L
  Day 57: number analyzed (Participants) | 17 | 12
  Day 57 | -0.32 (2.192) | -7.78 (27.500)
  Day 85: number analyzed (Participants) | 14 | 11
  Day 85 | -0.62 (2.180) | 0.24 (1.692)
  EOS: number analyzed (Participants) | 14 | 11
  EOS | 0.19 (3.432) | 0.05 (1.015)

12. Secondary Outcome: LYS006 Plasma Concentration
Description: LYS006 plasma concentrations were determined by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. No methods for imputation of missing data were used.
Time Frame: pre-dose at Days 1, 29, 57 and 85 and post-dose (1, 2, 3 and 4 hours) at Days 29 and 57
Population: The overall number of participants analyzed includes all participants. The number analyzed per row represents participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 21
ng / mL
  Day 1 (0 h): number analyzed (Participants) | 16 | 14
  Day 1 (0 h) | 0.162 (0.648) | 0.00 (0.00)
  Day 29 (0 h): number analyzed (Participants) | 7 | 7
  Day 29 (0 h) | 78.9 (74.0) | 53.5 (74.9)
  Day 29 (1 h): number analyzed (Participants) | 18 | 17
  Day 29 (1 h) | 174 (89.6) | 169 (105)
  Day 29 (2 h): number analyzed (Participants) | 18 | 18
  Day 29 (2 h) | 224 (113) | 189 (105)
  Day 29 (3 h): number analyzed (Participants) | 17 | 17
  Day 29 (3 h) | 188 (89.8) | 145 (54.9)
  Day 29 (4 h): number analyzed (Participants) | 18 | 16
  Day 29 (4 h) | 149 (73.6) | 110 (31.8)
  Day 57 (0 h): number analyzed (Participants) | 12 | 9
  Day 57 (0 h) | 58.0 (57.2) | 24.0 (21.4)
  Day 57 (1 h): number analyzed (Participants) | 16 | 13
  Day 57 (1 h) | 200 (118) | 123 (123)
  Day 57 (2 h): number analyzed (Participants) | 17 | 15
  Day 57 (2 h) | 222 (80.3) | 198 (88.7)
  Day 57 (3 h): number analyzed (Participants) | 17 | 15
  Day 57 (3 h) | 188 (74.3) | 156 (59.2)
  Day 57 (4 h): number analyzed (Participants) | 17 | 15
  Day 57 (4 h) | 140 (83.3) | 126 (54.1)
  Day 85 (0 h): number analyzed (Participants) | 7 | 4
  Day 85 (0 h) | 15.2 (17.6) | 10.2 (18.7)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of LYS006
Description: LYS006 plasma concentrations were determined by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. Cmax of LYS006 was determined with Phoenix WinNonlin (Version 8.0 or higher). No methods for imputation of missing data were used.
Time Frame: pre-dose and post-dose (1, 2, 3 and 4 hours) at Days 29 and 57
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | LYS006 | LYS006 + LJN452
Number analyzed (Participants) | 20 | 21
ng / mL
  Day 29: number analyzed (Participants) | 18 | 16
  Day 29 | 264 (87.7) | 215 (98.8)
  Day 57: number analyzed (Participants) | 17 | 15
  Day 57 | 271 (71.1) | 228 (88.1)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 113 days.
Description: Any sign or symptom that occurs during the study treatment plus the 28 days post treatment
Groups:
- Total: Total
Arm/Group | LYS006 | LYS006 + LJN452 | Total
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/41
Other Adverse Events (participants affected / at risk) | 9/20 | 15/21 | 24/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LYS006 (N=20) | LYS006 + LJN452 (N=21) | Total (N=41)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 2 | 5
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 4
Dizziness (Nervous system disorders) | 2 | 0 | 2
Headache (Nervous system disorders) | 4 | 4 | 8
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 13 | 13
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT04147195/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT04147195/SAP_001.pdf